CLINICAL TRIAL: NCT00337896
Title: T and B Cell Immune Responses to Influenza A/H5N1 Vaccine
Brief Title: T and B Cell Response to Avian Flu Vaccine
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 06-0005
Record Dates: First submitted 2006-06-15; First posted 2006-06-20 (Estimated); Last update posted 2013-08-16 (Estimated); Status verified 2011-04

CONDITIONS: Influenza
Keywords: vaccine, influenza, A/H5N1, CMI, sub-study
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood

GROUPS / COHORTS (1):
- observation: healthy adults ages 18-64 years, enrolled at Stanford University Hospital and participating in another clinical trial (DMID Protocol 04-062)

SUMMARY:
The purpose of this substudy study is to evaluate the types of cells involved in fighting infection to the A/H5N1 (avian flu virus) vaccine. A maximum of 30 healthy adults ages 18-64 years, enrolled at Stanford University Hospital and participating in another clinical trial (DMID Protocol 04-062) will be enrolled into this substudy to collect additional samples of blood for testing before and approximately one week after each vaccination.

DETAILED DESCRIPTION:
A human vaccination trial involving influenza A/H5N1 vaccine with different adjuvants is being conducted in a healthy adult population aged 18-64 years (DMID 04-062) to test the safety, reactogenicity, and immunogenicity of monovalent inactivated influenza A/H5N1 vaccine when given with either alone (no adjuvant), or given along with either alum or MF59. Two doses of the vaccine/adjuvent will be administered day 0 and day 28. This study is linked to DMID protocol 04-062. This protocol is a substudy to collect additional blood samples to specifically evaluate the cell-mediated immune responses generated from the vaccine. Primary goals of this study are 1) to establish reproducible, functional cell-mediate immune response assays to evaluate the magnitude and functional capacity of B cells, NK cells and T cells responding to monovalent subvirion H5 influenza vaccine 2) to evaluate the percent of subjects demonstrating B cell, NK cell, CD8+ and/or CD4+ response. The secondary goal of this study is to examine and compare the adjuvant effect of Alum or MF59 compared to no adjuvant on cell mediated immune responses.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects who are eligible and enrolled in 04-062 and have agreed to the extra blood draws for this substudy will be considered for enrollment if they will be receiving 15 micorgrams of the H5N1 vaccine without an adjuvant or with 15 micrograms of the H5N1 vaccine with alum or MF59 adjuvant. Subjects will not be recruited outside the main vaccine trial.
2. Subjects who understand and sign the consent form for this study.
3. Subjects who meet pre-screening qualifications will be eligible for the initial pre-vaccination blood draw.

Exclusion Criteria:

1. All subjects who are ineligible for the main monovalent subvirion H5 vaccine trials will not be eligible for the CMI sub-study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy adults male and female ages 18-64 years, participating in another clinical trial (DMID Protocol 04-062)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2006-03; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States